CLINICAL TRIAL: NCT02365402
Title: Efficacies of Entecavir Add on HBeAg Negative Chronic Hepatitis B Patients With HBV DNA Load ≥1000 Copies/ml After 3 Months of Peginterferon Alpha 2a Treatment
Brief Title: Efficacies of Entecavir Add on HBeAg Negative Patients With HBV DNA Positive During Peginterferon Alpha 2a Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, liver diseases center, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTXY006
Record Dates: First submitted 2015-02-15; First posted 2015-02-18 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; peginterferon; sustained viral response; entecavir; HBeAg
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- entecavir with PEG-IFN a-2a (Experimental): After enrolled, entecavir will added, and patients will receive treatment of PEG-IFN a-2a combine with entecavir for 48 weeks and 24 weeks of follow up after treatment.
  Interventions: Drug: Entecavir
- control group (No Intervention): In this group, patients will be continue treated only by PEG-IFN a-2a for 48 weeks after enrolled and receive 24 weeks of follow up.

INTERVENTIONS:
Drug: Entecavir — After enrolled, entecavir will added, and patients will receive treatment of PEG-IFN a-2a combine with entecavir for 48 weeks and 24 weeks of follow-up after treatment.
  Arms: entecavir with PEG-IFN a-2a

SUMMARY:
The aim of interferon therapy in HBeAg negative chronic hepatitis B was to make patients obtain immune control to hepatitis B virus defined as sustained viral response after treatment. However this target could not be get if patients keep HBV DNA positive during interferon treatment and offend relapse after treatment withdraw. In this trail, entecavir will add on patients with HBV DNA load ≥1000copies/ml after 3 months of peginterferon alpha 2a treatment, and the efficacies of the combine treatment will be evaluated by the rate of sustained viral response after 48 weeks of treatment and 24 week follow up.

DETAILED DESCRIPTION:
HBeAg negative patients with HBV DNA load ≥1000copies/ml after 3 months of peginterferon alpha 2a treatment would be randomize enrolled into two groups, in Interventional group, patients will receive entecavir combine with peginterferon alpha 2a treatment for 48 weeks and followed 24 weeks. Patients in control group will be continue treated only by peginterferon alpha 2a for 48 weeks and followed 24 weeks after treatment. Serum HBV DNA load, HBsAg/anti-HBs level, HBeAg/anti-HBe will be tested at enrollment and every 3 months during the treatment course. Parameters of Liver and kidney function, and liver ultrasound examination will be tested with intervals 1-3 months. The efficacies of combined therapy were evaluated by the rate of sustained viral response after 48 weeks treatment and 24 weeks follow up compared with control group.

ELIGIBILITY:
Inclusion Criteria:

* HBeAg negative patients with HBV DNA load ≥1000copies/ml after 3 months of peginterferon a-2a treatment

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
rate of sustained virual response | 72 weeks
  sustained viral response was defined as serum HBV DNA load was undetectable at the end of treatment and 24 weeks of follow-up.

SECONDARY OUTCOMES:
rates of HBsAg loss during treatment course and at the end of follow-up | 72 weeks
  HBsAg loss defined as HBsAg level ≤0.05 IU/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China